CLINICAL TRIAL: NCT05902780
Title: Can Caudal Dexmedetomidine Provide Effective Analgesia During Pediatric Inguinoscrotal Surgery?
Brief Title: Can Caudal Dexmedetomidine Provide Effective Analgesia?
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Nourhan Elsayed Mohamed Amer, Lecturer of Anesthesia at Faculty of Medicine, Benha University, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Dexmedetomidine
Record Dates: First submitted 2023-05-23; First posted 2023-06-15 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Anesthesia; Local Anesthesia
Keywords: Anesthesia; Caudal; Epidural; Regional; postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group B (25 patients) (Active Comparator): In this group, and after induction of general anesthesia, pediatric patients will receive a caudal injection of bupivacaine 0.125 % in a dose of 1ml/kg.
  Interventions: Drug: Caudal Bupivacaine injection
- Group D (25 patients) (Active Comparator): In this group, and after induction of general anesthesia, pediatric patients will receive a caudal injection of dexmedetomidine in a dose of 1.5 mcg/kg.
  Interventions: Drug: Caudal Dexmedetomidine Injection

INTERVENTIONS:
Drug: Caudal Bupivacaine injection — - Group B (n =25): In this group, and after induction of general anesthesia, pediatric patients will receive a caudal injection of bupivacaine 0.125 % in a dose of 1ml/kg.
  Arms: Group B (25 patients)
Drug: Caudal Dexmedetomidine Injection — - Group D (n =25): In this group, and after induction of general anesthesia, pediatric patients will receive a caudal injection of dexmedetomidine in a dose of 1.5 mcg/kg.
  Arms: Group D (25 patients)

SUMMARY:
The goal of this clinical trial is to evaluate if caudal dexmedetomidine can provide effective analgesia during inguinoscrotal surgeries in pediatrics, if used caudally alone (and not as an adjunct to caudal bupivacaine).

The main question it aims to answer is:

* Can caudal dexmedetomidine provide effective analgesia? Participants will be pediatrics aged from 1 to 6 years ASA-I and ASA-II undergoing inguinoscrotal surgeries.

  - A total of 50 pediatric patients who will undergo inguinoscrotal surgery will be allocated randomly into 2 equal groups:
* Group B (n =25): In this group, and after induction of general anesthesia, pediatric patients will receive a caudal injection of bupivacaine 0.125 % in a dose of 1ml/kg.
* Group D (n =25): In this group, and after injection of general anesthesia, pediatric patients will receive a caudal injection of dexmedetomidine in a dose of 1.5 mcg/kg.

DETAILED DESCRIPTION:
• Introduction

* Caudal anesthesia is a relatively low-risk technique commonly used, either on its own or in combination with sedation or general anesthesia.
* Caudal anesthesia is one of the most used-popular regional blocks in children. This technique is a useful adjunct during general anesthesia and for providing postoperative analgesia after infra-umbilical operations.
* Caudal blocks performed on sedated children, enable not only early ambulation, but also periprocedural hemodynamic stability and spontaneous breathing in patient groups at maximum risk of a difficult airway. These are important advantages over general anesthesia, notably in preterm babies and in children with cardiopulmonary co-morbidities. Caudal epidural anesthesia has been shown to reduce stress response and shorten the time for extubation in children.
* Caudal anesthesia is indicated for surgical and non-surgical painful interventions in body areas from the sub-umbilical region downwards. Examples include procedures such as inguinal hernia repair, cystoscopy/transurethral manipulation, circumcision, anal atresia, treatment of limb ischemia, treatment of intussusception, or cast application to immobilize newborns with hip dysplasia.
* Contraindications to caudal anesthesia in children would include local site infection, pilonidal cyst, or spinal dysraphism such as tethered cord syndrome.
* Bupivacaine (an amide local anesthetic) has provided reliable anesthesia and analgesia.
* Bupivacaine is the indicated local anesthetic in caudal, epidural, and spinal anesthesia and is widely used clinically to manage acute and chronic pain. In addition to blocking Na+ channels, bupivacaine affects the activity of many other channels, including NMDA receptors.
* Adverse effects of bupivacaine includes local anesthetic systemic toxicity, urinary retention, high block, hypotension, delayed respiratory depression, and cardiac arrest.
* Dexmedetomidine is an alpha agonist having sedative, anxiolytic, hypnotic, analgesic, and sympatholytic properties. It produces these effects by inhibiting central sympathetic outflow by blocking the alpha receptors in the brainstem, thereby inhibiting the release of norepinephrine.
* Dexmedetomidine is a highly selective α2-adrenergic receptor agonist, which binds to transmembrane G protein-binding adrenoreceptors in the periphery (α2A), brain, and spinal cord (α2B, α2C) tissues.

In contrast to other sedative agents, dexmedetomidine, by acting on α2 receptors in the locus caeruleus, has potential analgesic effects without respiratory depression.

* Dexmedetomidine seems to help to reduce the time for extubation.
* Dexmedetomidine is also an adjunct infusion during general anesthesia. There is evidence that dexmedetomidine decreases postoperative pain, postoperative opioid usage, and nausea. This effect has also been shown to be present when using dexmedetomidine for sedation during procedures performed under spinal anesthesia. There has been some interest in using dexmedetomidine as an adjunct to prevent emergence agitation, postoperative delirium, and postoperative cognitive dysfunction. There is evidence for the prevention of emergence agitation in both children and adults.
* The most common adverse effects of dexmedetomidine are hypotension and bradycardia which result from the stimulation of presynaptic alpha receptors, which leads to a decreased release of norepinephrine; this is in addition to the decrease in the central sympathetic outflow. These are concerns regardless of the route of administration.

Ethical consideration :

The study protocol will be approved by the Institutional Research Ethics Committee. Informed written consent will be obtained from all parents of the pediatric patients, after being explained the purpose of the study and will be ensured strict confidentiality. They will be given the option of not participating in the study if they do not want to.

Type and design of the study:

• Study population: The study will be conducted at Benha University Surgical Hospital starting from July 2023 on pediatrics aged from 1 to 6 years ASA-I and ASA-II undergoing inguinoscrotal surgeries.

• Study design: Randomized prospective single-blind study.

* Sample size calculation The sample size was calculated using Power and Sample Size software version 3 based on a previous study, which explore the analgesic effect of caudal dexmedetomidine versus caudal morphine if used as an adjunct to bupivacaine in pediatric infra-umbilical surgery. The total sample size calculated was 50 patients (25 patients in each group).
* Methods:

A total of 50 pediatric patients who will undergo inguinoscrotal surgery will be allocated randomly into 2 equal groups:

Group B (n =25): In this group, and after induction of general anesthesia, pediatric patients will receive a caudal injection of bupivacaine 0.125 % in a dose of 1ml/kg Group D (n =25): In this group, and after induction of general anesthesia, pediatric patients will receive a caudal injection of dexmedetomidine in a dose of 1.5 mcg/kg.

• Aim of the work: The main objective of our study is to evaluate if caudal dexmedetomidine can provide effective analgesia during inguinoscrotal surgeries in pediatrics.

ELIGIBILITY:
Inclusion Criteria:

* ASA-I and ASA-II pediatric patients (age :1-6 years old)
* Inguinoscrotal surgeries

Exclusion Criteria:

* Patient's parent's refusal
* Unable to give consent
* Known allergy to the study medications
* Coagulopathies or on anticoagulant medications
* ASA-III or ASA-IV

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Amount of opioids needed by patients. | Intraoperative (during the surgery)
  How much opioids in mcg/kg will the patient needs
Amount of opioids needed by patients. | during the first 6 hours postoperative
  How much opioids in mcg/kg will the patient needs
Time to the first analgesic rescue | during the first 6 hours postoperative
  Measure time in minutes (min) till the patient needs opioids for the first time postoperative

SECONDARY OUTCOMES:
Blood pressure | Preoperative,Intraoperative and 2 hours postoperative
  Measure blood pressure in mmHg of the patient every 10 min
Heart rate | Preoperative, intraoperative, and 2 hours postoperative
  Measure heart rate in beat/min every 10 min
Emergence agitation | Intraoperative with extubation
  The incidence of emergence agitation is high in children, the level of agitation will be assessed through Paediatric Anesthesia Emergence Delirium Scale (PAED SCALE) which consist of 5 criteria that are scored using 5-point scale. The scores of each criterion are added to make a total score. The maximum achieved score is 20.
Presence of respiratory depression | 2 hours Postoperative every 10 min
  Measure respiratory rate in breath/ min